CLINICAL TRIAL: NCT01190215
Title: Immunogenicity and Safety Study of GSK Biologicals' Seasonal (2010-2011) Influenza Vaccine FluarixTM in Adolescents Previously Vaccinated With GSK Biologicals' H1N1 Vaccine PandemrixTM
Brief Title: Immunogenicity and Safety Study of FluarixTM Vaccine in Children Who Have Previously Been Vaccinated With PandemrixTM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 114452
Record Dates: First submitted 2010-08-26; First posted 2010-08-27 (Estimated); Results first posted 2012-07-13 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2017-08

CONDITIONS: Influenza
Keywords: Influenza; Pandemrix; H1N1; Fluarix
MeSH Terms: conditions — Influenza, Human

ARMS (2):
- Fluarix Group (Experimental): Subjects previously vaccinated with Pandemrix vaccine received 1 dose of Fluarix vaccine. All vaccines were administered in the deltoid region of the non-dominant arm on Day 0.
  Interventions: Biological: FluarixTM
- Havrix Group (Active Comparator): Subjects previously vaccinated with Pandemrix vaccine received 1 first dose of Havrix vaccine (subjects aged above 15 years) or Havrix-Junior vaccine (subjects aged 15 years and below). A second dose was given outside the study setting, at Month 6. All vaccines were administered in the deltoid region of the non-dominant arm on Day 0.
  Interventions: Biological: HavrixTM Junior (in subjects of 15 years old or below) or HavrixTM (in subjects above 15 years old)

INTERVENTIONS:
Biological: FluarixTM — One Intramuscular injection
  Arms: Fluarix Group
Biological: HavrixTM Junior (in subjects of 15 years old or below) or HavrixTM (in subjects above 15 years old) — Two Intramuscular injections
  Arms: Havrix Group

SUMMARY:
This study is designed to assess the immunogenicity, reactogenicity and safety following vaccination with GSK Biologicals' FluarixTM vaccine in children who have previously been vaccinated with one dose of PandemrixTM at the age of 10-17 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having previously been immunized with only one single dose of Pandemrix at the age of 10-17 years inclusive.
* Subjects having received Pandemrix at least six months prior to study enrolment.
* Subjects who the investigator believes that subject and/or parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol
* Written informed consent obtained from the subject/ the parent(s)/LAR(s) of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects or Parent(s)/LAR(s) with access to a consistent means of telephone contact, land line or mobile, but NOT a pay phone or other multiple-user device

Exclusion Criteria:

* Active participation in other clinical trials.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccine or planned use during the study period.
* Planned administration of any vaccine 30 days prior and 30 days after any study vaccine administration.
* Chronic administration of immunosuppressants or other immune-modifying drugs within three months prior to enrolment in this study or planned administration during the study period.
* Acute disease and/or fever at the time of enrolment:
* Acute or chronic, clinically-significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history and physical examination.
* Administration of immunoglobulins and/or any blood products within the three months prior to the enrolment in this study, or planned use during the study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* History of seizures or progressive neurological disease.
* Subjects having received an H1N1v pandemic vaccine other than Pandemrix or having received the 2010/2011 seasonal influenza vaccine.
* If the subject is female and if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for two months after completion of the vaccination series.
* Child in care.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2010-10-04; Primary Completion 2011-07-07 (Actual); Study Completion 2011-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Vesikari T, Richardus JH, Berglund J, Korhonen T, Flodmark CE, Lindstrand A, Silfverdal SA, Bambure V, Caplanusi A, Dieussaert I, Roy-Ghanta S, Vaughn DW. Immunogenicity and Safety of a Trivalent Inactivated Influenza Vaccine in Children 6 Months to 17 Years of Age, Previously Vaccinated with an AS03-Adjuvanted A(H1N1)Pdm09 Vaccine: Two Open-label, Randomized Trials. Pediatr Infect Dis J. 2015 Jul;34(7):774-82. doi: 10.1097/INF.0000000000000709. PMID 26069949
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 114452 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114452 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114452 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114452 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114452 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114452 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Up to Day 28
Arm/Group | Fluarix Group | Havrix Group
Started | 38 | 39
Completed | 38 | 39
Not Completed | 0 | 0
Period: Up to Month 6
Arm/Group | Fluarix Group | Havrix Group
Started | 38 | 39
Completed | 36 | 39
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluarix Group | Havrix Group | Total
Number analyzed (Participants) | 38 | 39 | 77
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.6 (2.22) | 14.7 (2.28) | 14.7 (2.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 16 | 20 | 36

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Antibody Titres for Haemagglutination Inhibition (HI) Antibodies Against Fluarix Vaccine Containing H1N1 Strain.
Description: Fluarix vaccine strain was Flu A/California/7/2009 (H1N1).
  Day 28 data were presented only for the Fluarix Group.
  Titres were expressed as geometric mean antibody titre.
Time Frame: At Day 0 and Day 28
Population: The According-To-Protocol cohort for immunogenicity at Day 28 included subjects who received at least 1 vaccine dose, for whom data concerning immunogenicity outcome measures were available. It included subjects for whom assay results were available for antibodies against H1N1 antigen for the blood sample taken 28 days after the vaccine dose.
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 33 | 39
Titres
  Flu A/Cal/7/09 H1N1 [Day 0] | 150.1 [105.8 to 213.0] | 150.3 [106.0 to 213.3]
  Flu A/Cal/7/09 H1N1 [Day 28] | 646.8 [534.6 to 782.6] | NA [NA to NA] — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.

2. Primary Outcome: Number of Seropositive Subjects for Haemagglutination Inhibition (HI) Antibodies Against Fluarix Vaccine Containing H1N1 Strain.
Description: Fluarix vaccine strain was Flu A/California/7/2009 (H1N1).
  Seropositivity was assessed for subjects with an antibody titre assay cut-off value equal to or above 1:10.
  Day 28 data was presented only for the Fluarix Group.
Time Frame: At Day 0 and Day 28
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 33 | 39
Subjects
  Flu A/Cal/7/09 H1N1 [Day 0] | 33 | 39
  Flu A/Cal/7/09 H1N1 [Day 28] | 33 | NA — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.

3. Primary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against Fluarix Vaccine Containing H1N1 Strain.
Description: Fluarix vaccine strain was Flu A/California/7/2009 (H1N1).
  A seroconverted subject was a subject who had either a pre-vaccination (Day 0) titre less than (< ) 1:10 and a post-vaccination titre greater than or equal to ( ≥) 1:40 or a pre-vaccination titre ≥ 1:10 and at least a 4-fold increase in post-vaccination titre.
  Day 28 data were presented for the Fluarix Group only.
Time Frame: At Day 28
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 33 | 0
Subjects | 16 |

4. Primary Outcome: Number of Seroprotected Subjects for Haemagglutination Inhibition (HI) Antibodies Against Fluarix Vaccine Containing H1N1 Strain.
Description: Fluarix vaccine strain was Flu A/California/7/2009 (H1N1).
  A seroprotected subject was a subject with a serum HI titre ≥ 1:40 that usually is accepted as indicating protection.
  Day 28 data were presented for the Fluarix Group only.
Time Frame: At Day 0 and Day 28
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 33 | 39
Subjects
  Flu A/Cal/7/09 H1N1 [Day 0] | 31 | 36
  Flu A/Cal/7/09 H1N1 [Day 28] | 33 | NA — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.

5. Primary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibodies Against Fluarix Vaccine Containing H1N1 Strain.
Description: Fluarix vaccine strain was Flu A/California/7/2009 (H1N1).
  MGI is defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titre to the pre-vaccination (Day 0) reciprocal HI titre.
  Day 28 data were presented for the Fluarix Group only.
Time Frame: At Day 28
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 33 | 0
Ratio | 4.3 [2.9 to 6.4] |

6. Secondary Outcome: Geometric Mean Antibody Titres for Haemagglutination Inhibition (HI) Antibodies Against All Fluarix Vaccine Strains.
Description: Fluarix vaccine strains were Flu A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2) and B/Brisbane/60/2008.
  Day 28 data were presented for the Fluarix Group only.
  Titres were expressed as geometric mean antibody titres (GMTs).
Time Frame: At Day 0 and Day 28
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 33 | 39
Titres
  Flu A/Cal/7/09 H1N1 [Day 0] | 150.1 [105.8 to 213.0] | 150.3 [106.0 to 213.3]
  Flu A/Cal/7/09 H1N1 [Day 28] | 646.8 [534.6 to 782.6] | NA [NA to NA] — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.
  Flu B/Bri/60/08 Victoria [Day 0] | 22.2 [14.7 to 33.5] | 21.0 [14.8 to 30.0]
  Flu B/Bri/60/08 Victoria [Day 28] | 320.1 [216.8 to 472.6] | NA [NA to NA] — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.
  Flu A/Vic/210/09 H3N2 [Day 0] | 20.0 [13.0 to 30.8] | 279.2 [202.1 to 385.8]
  Flu A/Vic/210/09 H3N2 [Day 28] | 20.3 [13.9 to 29.8] | NA [NA to NA] — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.

7. Secondary Outcome: Geometric Mean Antibody Titres for Haemagglutination Inhibition (HI) Antibodies Against All Fluarix Vaccine Strains.
Description: Fluarix vaccine strains were Flu A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2) and B/Brisbane/60/2008.
  Only data for the Flu A/California/7/2009 (H1N1) strain were presented for the Havrix Group.
  Titres were expressed as geometric mean antibody titres (GMTs).
Time Frame: At Day 0 and at Month 6
Population: Analysis was performed on According-to-Protocol (ATP) cohort for antibody persistence at Month 6 which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available at Month 6.
Measure: Geometric Mean (95% Confidence Interval); unit: Titres
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 35 | 37
Titres
  Flu B/Bri/60/08 Victoria [Day 0] | 22.9 [15.6 to 33.8] | NA [NA to NA] — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu B/Bri/60/08 Victoria [Month 6] | 242.4 [173.9 to 337.8] | NA [NA to NA] — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu A/Cal/7/09 H1N1 [Day 0] | 169.7 [116.2 to 247.8] | 152.7 [105.6 to 220.8]
  Flu A/Cal/7/09 H1N1 [Month 6] | 346.4 [273.4 to 438.8] | 131.4 [92.5 to 186.6]
  Flu A/Vic/210/09 H3N2 [Day 0] | 17.9 [12.7 to 25.3] | NA [NA to NA] — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu A/Vic/210/09 H3N2 [Month 6] | 160.1 [118.1 to 217.0] | NA [NA to NA] — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.

8. Secondary Outcome: Number of Seropositive Subjects for Haemagglutination Inhibition (HI) Antibodies Against All Fluarix Vaccine Strains.
Description: Fluarix vaccine strains were Flu A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2) and B/Brisbane/60/2008.
  Seropositivity was assessed for subjects with an antibody titre assay cut-off value equal to or above 1:10.
  Day 28 data were presented for the Fluarix Group only.
Time Frame: At Day 0 and Day 28
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 33 | 39
Subjects
  Flu A/Cal/7/09 H1N1 [Day 0] | 33 | 39
  Flu A/Cal/7/09 H1N1 [Day 28] | 33 | NA — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.
  Flu B/Bri/60/08 Victoria [Day 0] | 26 | 31
  Flu B/Bri/60/08 Victoria [Day 28] | 33 | NA — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.
  Flu A/Vic/210/09 H3N2 [Day 0] | 24 | 28
  Flu A/Vic/210/09 H3N2 [Day 28] | 33 | NA — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.

9. Secondary Outcome: Number of Seropositive Subjects for Haemagglutination Inhibition (HI) Antibodies Against All Fluarix Vaccine Strains.
Description: Fluarix vaccine strains were Flu A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2) and B/Brisbane/60/2008.
  Seropositivity was assessed for subjects with an antibody titre assay cut-off equal to or above 1:10.
  Only data for the Flu A/California/7/2009 (H1N1) strain were presented for the Havrix Group.
Time Frame: At Day 0 and at Month 6
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 35 | 37
Subjects
  Flu B/Bri/60/08 Victoria [Day 0] | 29 | NA — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu B/Bri/60/08 Victoria [Month 6] | 35 | NA — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu A/Cal/7/09 H1N1 [Day 0] | 35 | 37
  Flu A/Cal/7/09 H1N1 [Month 6] | 35 | 37
  Flu A/Vic/210/09 H3N2 [Day 0] | 25 | NA — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu A/Vic/210/09 H3N2 [Month 6] | 35 | NA — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.

10. Secondary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against All Fluarix Vaccine Strains.
Description: Fluarix vaccine strains were Flu A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2) and B/Brisbane/60/2008.
  A seroconverted subject was a subject who had either a pre-vaccination (Day 0) titre less than (< ) 1:10 and a post-vaccination titre greater than or equal to ( ≥) 1:40 or a pre-vaccination titre ≥ 1:10 and at least a 4-fold increase in post-vaccination titre.
  Day 28 data were presented for the Fluarix Group only.
Time Frame: At Day 28
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 33 | 0
Subjects
  Flu A/Cal/7/09 H1N1 | 16 |
  Flu B/Bri/60/08 Victoria | 28 |
  Flu A/Vic/210/09 H3N2 | 29 |

11. Secondary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against All Fluarix Vaccine Strains.
Description: Fluarix vaccine strains were Flu A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2) and B/Brisbane/60/2008.
  A seroconverted subject was a subject who had either a pre-vaccination (Day 0) titre < 1:10 and a post-vaccination titre ≥ 1:40 or a pre-vaccination titre ≥ 1:10 and at least a 4-fold increase in post-vaccination titre.
  Only data for the Flu A/California/7/2009 (H1N1) strain were presented for the Havrix Group.
Time Frame: At Month 6
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 35 | 37
Subjects
  Flu B/Bri/60/08 Victoria | 29 | NA — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu A/Cal/7/09 H1N1 | 8 | 2
  Flu A/Vic/210/09 H3N2 | 30 | NA — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.

12. Secondary Outcome: Number of Seroprotected Subjects for Haemagglutination Inhibition (HI) Antibodies Against All Fluarix Vaccine Strains.
Description: Fluarix vaccine strains were Flu A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2) and B/Brisbane/60/2008.
  A seroprotected subject was a subject with a serum HI titre ≥ 1:40 that usually is accepted as indicating protection.
  Day 28 data were presented for the Fluarix Group only.
Time Frame: At Day 0 and Day 28
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 33 | 39
Subjects
  Flu A/Cal/7/09 H1N1 [Day 0] | 31 | 36
  Flu A/Cal/7/09 H1N1 [Day 28] | 33 | NA — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.
  Flu B/Bri/60/08 Victoria [Day 0] | 13 | 11
  Flu B/Bri/60/08 Victoria [Day 28] | 33 | NA — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.
  Flu A/Vic/210/09 H3N2 [Day 0] | 12 | 16
  Flu A/Vic/210/09 H3N2 [Day 28] | 33 | NA — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.

13. Secondary Outcome: Number of Seroprotected Subjects for Haemagglutination Inhibition (HI) Antibodies Against All Fluarix Vaccine Strains.
Description: Fluarix vaccine strains were Flu A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2) and B/Brisbane/60/2008.
  A seroprotected subject was a subject with a serum HI titre ≥ 1:40 that usually is accepted as indicating protection.
  Only data for the Flu A/California/7/2009 (H1N1) strain were presented for the Havrix Group.
Time Frame: At Day 0 and Month 6
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 35 | 37
Subjects
  Flu B/Bri/60/08 Victoria [Day 0] | 13 | NA — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu B/Bri/60/08 Victoria [Month 6] | 33 | NA — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu A/Cal/7/09 H1N1 [Day 0] | 33 | 34
  Flu A/Cal/7/09 H1N1 [Month 6] | 35 | 34
  Flu A/Vic/210/09 H3N2 [Day 0] | 13 | NA — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu A/Vic/210/09 H3N2 [Month 6] | 34 | NA — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.

14. Secondary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibodies Against All Fluarix Vaccine Strains.
Description: Fluarix vaccine strains were Flu A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2) and B/Brisbane/60/2008.
  MGI is defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titre to the pre-vaccination (Day 0) reciprocal HI titre.
  Day 28 data were presented for the Fluarix Group only.
Time Frame: At Day 28
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 33 | 0
Ratio
  Flu A/Cal/7/09 H1N1 | 4.3 [2.9 to 6.4] |
  Flu B/Bri/60/08 Victoria | 14.4 [9.4 to 22.0] |
  Flu A/Vic/210/09 H3N2 | 14.0 [9.3 to 21.1] |

15. Secondary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibodies Against All Fluarix Vaccine Strains.
Description: Fluarix vaccine strains were Flu A/California/7/2009 (H1N1), A/Victoria/210/2009 (H3N2) and B/Brisbane/60/2008.
  MGI is defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titre to the pre-vaccination (Day 0) reciprocal HI titre.
  Only data for the Flu A/California/7/2009 (H1N1) strain were presented for the Havrix Group.
Time Frame: At Month 6
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 35 | 37
Ratio
  Flu B/Bri/60/08 Victoria | 10.6 [7.5 to 14.9] | NA [NA to NA] — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu A/Cal/7/09 H1N1 | 2.0 [1.6 to 2.7] | 0.9 [0.7 to 1.1]
  Flu A/Vic/210/09 H3N2 | 8.9 [6.6 to 12.0] | NA [NA to NA] — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.

16. Secondary Outcome: Geometric Mean Antibody Titres for Neutralising Antibodies Against All Fluarix Vaccine Strains.
Description: Fluarix vaccine strains were Flu A/California/7/2009 (H1N1), A/Perth/16/09(H3N2) and B/Brisbane/60/2008.
  Day 28 data were presented for the Fluarix Group only.
  Titres were expressed as geometric mean antibody titres (GMTs).
Time Frame: At Day 0 and at Day 28
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titre
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 33 | 39
titre
  Flu B/Bri/60/08 Victoria [Day 0] | 26.0 [20.2 to 33.6] | 24.5 [18.9 to 31.9]
  Flu B/Bri/60/08 Victoria [Day 28] | 257.9 [158.5 to 419.5] | NA [NA to NA] — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.
  Flu A/Cal/7/09 H1N1 [Day 0] | 119.7 [95.2 to 150.5] | 137.7 [108.0 to 175.5]
  Flu A/Cal/7/09 H1N1 [Day 28] | 1512.4 [1077.9 to 2122.1] | NA [NA to NA] — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.
  Flu A/Per/16/09 H3N2 [Day 0] | 69.8 [50.5 to 96.5] | 72.6 [55.2 to 95.5]
  Flu A/Per/16/09 H3N2 [Day 28] | 614.5 [371.4 to 1016.7] | NA [NA to NA] — No blood samples were collected at Day 28 on subjects from the Havrix Group for antibody determination.

17. Secondary Outcome: Geometric Mean Antibody Titres for Neutralising Antibodies Against All Fluarix Vaccine Strains.
Description: Fluarix vaccine strains were Flu A/California/7/2009 (H1N1), A/Perth/16/09 (H3N2) and B/Brisbane/60/2008.
  Titres were expressed as geometric mean antibody titres (GMTs).
Time Frame: At Day 0 and at Month 6
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: titre
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 35 | 37
titre
  Flu B/Bri/60/08 Victoria [Day 0] | 25.1 [19.7 to 32.1] | NA [NA to NA] — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu B/Bri/60/08 Victoria [Month 6] | 199.5 [145.8 to 273.0] | NA [NA to NA] — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu A/Cal/7/09 H1N1 [Day 0] | 119.4 [94.5 to 150.8] | 138.3 [107.5 to 178.0]
  Flu A/Cal/7/09 H1N1 [Month 6] | 390.6 [291.4 to 523.8] | 115.3 [82.4 to 161.4]
  Flu A/Per/16/09 H3N2 [Day 0] | 62.5 [49.5 to 78.8] | NA [NA to NA] — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu A/Per/16/09 H3N2 [Month 6] | 266.8 [173.6 to 410.1] | NA [NA to NA] — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.

18. Secondary Outcome: Number of Seroconverted Subjects for Neutralising Antibodies Against All Fluarix Vaccine Strains.
Description: A seroconverted subject for neutralising antibodies was a subject with a minimum 4-fold increase in titre at post-vaccination.
  Fluarix vaccine strains were Flu A/California/7/2009 (H1N1), A/Perth/16/09 (H3N2) and B/Brisbane/60/2008.
  Day 28 data were presented for the Fluarix Group only.
Time Frame: At Day 28
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 33 | 0
Subjects
  Flu B/Bri/60/08 Victoria | 25 |
  Flu A/Cal/7/09 H1N1 | 29 |
  Flu A/Per/16/09 H3N2 | 22 |

19. Secondary Outcome: Number of Seroconverted Subjects for Neutralising Antibodies Against All Fluarix Vaccine Strains.
Description: A seroconverted subject for neutralising antibodies was a subject with a minimum 4-fold increase in titre at post-vaccination.
  Fluarix vaccine strains were Flu A/California/7/2009 (H1N1), A/Perth/16/09 (H3N2) and B/Brisbane/60/2008.
  At Month 6, only data for the Flu A/California/7/2009 (H1N1) strain were presented for the Havrix Group.
Time Frame: At Month 6
Population: as for outcome 7
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 35 | 37
Subjects
  Flu B/Bri/60/08 Victoria | 28 | NA — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.
  Flu A/Cal/7/09 H1N1 | 13 | 2
  Flu A/Per/16/09 H3N2 | 17 | NA — Data for Havrix Group was presented only for the Flu A/California/7/2009 (H1N1) strain as per protocol.

20. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of any solicited local symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling above 50 millimetres.
Time Frame: Within 7 days (Day 0 - Day 6) after vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 38 | 39
Subjects
  Any pain | 35 | 24
  Grade 3 pain | 2 | 0
  Any redness | 6 | 5
  Grade 3 redness | 0 | 0
  Any swelling | 5 | 0
  Grade 3 swelling | 1 | 0

21. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited General Symptoms.
Description: Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, shivering, sweating, temperature (temperature = axillary temperature equal to or above 37.5 degrees Celsius).
  Any = occurrence of any solicited general symptom regardless of intensity grade or relation to vaccination. Grade 3 symptom = general symptom that prevented normal activity. Grade 3 temperature = axillary temperature above 39.0 degrees Celsius.
Time Frame: Within 7 days (Day 0 - Day 6) after vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 38 | 39
Subjects
  Any arthralgia | 4 | 5
  Grade 3 arthralgia | 0 | 0
  Any fatigue | 25 | 24
  Grade 3 fatigue | 1 | 1
  Any gastrointestinal symptoms | 8 | 3
  Grade 3 gastrointestinal symptoms | 2 | 0
  Any headache | 24 | 16
  Grade 3 headache | 1 | 0
  Any myalgia | 16 | 16
  Grade 3 myalgia | 0 | 1
  Any shivering | 18 | 9
  Grade 3 shivering | 0 | 0
  Any sweating | 9 | 4
  Grade 3 sweating | 0 | 0
  Any temperature >= 37.5°C | 4 | 1
  Grade 3 temperature > 39.0°C | 0 | 0

22. Secondary Outcome: Number of Days With Any Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling.
  Inter-quartile range assessed was the 25th percentile and the 75th percentile.
Time Frame: Within 7 days (Day 0 - Day 6) after vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 38 | 39
Days
  Pain | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.5]
  Redness | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Swelling | 2.0 [2.0 to 3.0] | 0 [0 to 0]

23. Secondary Outcome: Number of Days With Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain and swelling.
  Grade 3 redness/swelling = redness/swelling above 50 millimetres.
  Inter-quartile range assessed was the 25th percentile and the 75th percentile.
Time Frame: Within 7 days (Day 0 - Day 6) after vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 38 | 39
Days
  Pain | 1.0 [1.0 to 1.0] | 0 [0 to 0]
  Swelling | 1.0 [1.0 to 1.0] | 0 [0 to 0]

24. Secondary Outcome: Number of Days With Any Solicited General Symptoms.
Description: Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, shivering, sweating, temperature (temperature = axillary temperature equal to or above 37.5 degrees Celsius).
  Inter-quartile range assessed was the 25th percentile and the 75th percentile.
Time Frame: Within 7 days (Day 0 - Day 6) after vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 38 | 39
Days
  Arthralgia | 2.0 [1.5 to 4.0] | 1.0 [1.0 to 2.0]
  Fatigue | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0]
  Gastrointestinal | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 3.0]
  Headache | 2.0 [1. to 3.0] | 1.0 [1.0 to 2.0]
  Myalgia | 2.0 [1.5 to 3.5] | 2.0 [1.0 to 3.0]
  Sweating | 1.0 [1.0 to 1.0] | 2.0 [2.0 to 2.5]
  Shivering | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 1.0]
  Temperature | 1.0 [1.0 to 1.5] | 1.0 [1.0 to 1.0]

25. Secondary Outcome: Number of Days With Grade 3 Solicited General Symptoms.
Description: Solicited general symptoms assessed were fatigue, gastrointestinal symptoms, headache and myalgia.
  Grade 3 symptom = general symptom that prevented normal activity.
  Inter-quartile range assessed was the 25th percentile and the 75th percentile.
Time Frame: Within 7 days (Day 0 - Day 6) after vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 38 | 39
Days
  Fatigue | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Gastrointestinal | 1.0 [1.0 to 1.0] | 0 [0 to 0]
  Headache | 1.0 [1.0 to 1.0] | 0 [0 to 0]
  Myalgia | 0 [0 to 0] | 1.0 [1.0 to 1.0]

26. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
  Grade 3 = event that prevented normal, everyday activities. Related = event assessed by the investigator as causally related to the study vaccination.
Time Frame: Within 28 days (Day 0 - Day 27) after vaccination
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 38 | 39
Subjects
  Any | 12 | 11
  Grade 3 | 1 | 2
  Related to vaccination | 4 | 1

27. Secondary Outcome: Number of Subjects Reporting Medically-attended Events (MAEs).
Description: For each solicited and unsolicited symptom the subject experienced, the subject was asked if they received medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel for any reason.
Time Frame: Within the 28-day (Days 0-27) post-vaccination period
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 38 | 39
Subjects | 1 | 3

28. Secondary Outcome: Number of Subjects Reporting Medically-attended Events (MAEs).
Description: as for outcome 27
Time Frame: During the entire study period (Up to Month 6)
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 38 | 39
Subjects | 2 | 4

29. Secondary Outcome: Number of Subjects Reporting Adverse Events of Specific Interest (AESIs)/Potential Immune Mediated Diseases (pIMDs).
Description: Potential Immune-Mediated Diseases (pIMDs) or Adverse events of specific interest (AESI), are a subset of AEs that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology.
Time Frame: During the entire study period (Up to Month 6)
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 38 | 39
Subjects | 0 | 0

30. Secondary Outcome: Number of Subjects Reporting Adverse Events of Special Interest.
Description: Adverse events of special interest for safety monitoring includes both convulsion and anaphylaxis.
Time Frame: During the entire study period (Up to Month 6)
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 38 | 39
Subjects | 0 | 0

31. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: Within the 28-day (Days 0-27) post-vaccination period
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 38 | 39
Subjects | 0 | 0

32. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs).
Description: as for outcome 31
Time Frame: During the entire study period (Up to Month 6)
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | Fluarix Group | Havrix Group
Number analyzed (Participants) | 38 | 39
Subjects | 1 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed up to Day 28 and during the entire study period, up to Month 6. Systematically and non-systematically assessed frequent adverse events were assessed during the 7 day and 28 day post-vaccination period respectively.
Arm/Group | Fluarix Group | Havrix Group
Serious Adverse Events (participants affected / at risk) | 1/38 | 0/39
Other Adverse Events (participants affected / at risk) | 37/38 | 34/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix Group (N=38) | Havrix Group (N=39)
Acute tonsillitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix Group (N=38) | Havrix Group (N=39)
Upper respiratory tract infection (Infections and infestations) | 3 | 2
Headache (Nervous system disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain (General disorders) | 35 | 24
Redness (General disorders) | 6 | 5
Swelling (General disorders) | 5 | 0
Arthralgia (General disorders) | 4 | 5
Fatigue (General disorders) | 25 | 24
Gastrointestinal symptoms (General disorders) | 8 | 3
Headache (General disorders) | 24 | 16
Myalgia (General disorders) | 16 | 16
Shivering (General disorders) | 18 | 9
Sweating (General disorders) | 9 | 4
Temperature (General disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.